CLINICAL TRIAL: NCT03324373
Title: Proof of Concept for Lenvatinib and Everolimus Prior to Nephrectomy in Eligible Patients With Local and Metastatic Renal Cell Carcinoma (RCC)
Brief Title: Lenvatinib and Everolimus in Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yousef Zakharia (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor-Investigator, Yousef Zakharia, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201710801
Record Dates: First submitted 2017-10-20; First posted 2017-10-27 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — lenvatinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenvatinib and Everolimus prior to cytoreductive nephrectomy (Experimental): Eligible patients will start treatment with lenvatinib 18 mg PO daily (administered as one 10 mg capsule and two 4 mg capsules) and everolimus 5 mg PO daily for 4 weeks constituting one cycle. Two cycles of treatment will be administered and after 2 weeks wash out period, the patients will go for nephrectomy.
  Interventions: Drug: Lenvatinib; Drug: Everolimus; Procedure: Partial or Radical Cytoreductive Nephrectomy

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib is a receptor tyrosine kinase (RTK) inhibitor that inhibits the kinase activities of vascular endothelial growth factor (VEGF) receptors VEGFR1 (FLT1), VEGFR2 (KDR), and VEGFR3 (FLT4). Lenvatinib also inhibits other RTKs that have been implicated in pathogenic angiogenesis, tumor growth, and cancer progression in addition to their normal cellular functions, including fibroblast growth factor (FGF) receptors FGFR1, 2, 3, and 4; the platelet derived growth factor receptor alpha (PDGFRα), KIT, and RET.
  Other Names: LENVIMA®, KISPLYX®
Drug: Everolimus — Everolimus is an inhibitor of mammalian target of rapamycin (mTOR), a serine-threonine kinase, downstream of the PI3K/AKT pathway. The mTOR pathway is dysregulated in several human cancers. Everolimus binds to an intracellular protein, FKBP-12, resulting in an inhibitory complex formation (mTORC1) and thus inhibition of mTOR kinase activity. Everolimus reduced the activity of S6 ribosomal protein kinase (S6K1) and eukaryotic elongation factor 4E-binding protein (4E-BP1), downstream effectors of mTOR, involved in protein synthesis. In addition, everolimus inhibited the expression of hypoxia-inducible factor (e.g., HIF-1) and reduced the expression of vascular endothelial growth factor (VEGF). Inhibition of mTOR by everolimus has been shown to reduce cell proliferation, angiogenesis, and glucose uptake in in vitro and/or in vivo studies.
  Other Names: AFINITOR®
Procedure: Partial or Radical Cytoreductive Nephrectomy — Surgical removal of a kidney.
  After completion of 8 weeks of therapy and restaging, investigators will require 2 weeks wash out period. The patients will be evaluated by urology oncology team and appropriate surgery will be planned. This includes partial nephrectomy and radical nephrectomy.

SUMMARY:
The purpose of this research study is to see what effect the combination of lenvatinib plus everolimus has in local and metastatic renal cell carcinoma to potentially make surgically unresectable tumors resectable.

DETAILED DESCRIPTION:
This is a pilot interventional clinical trial at the University of Iowa Hospitals and Clinics, enrolling 15 subjects and lasting approximately 12 months. Eligible patients will start treatment with lenvatinib 18 mg PO daily (administered as one 10 mg capsule and two 4 mg capsules) and everolimus 5 mg PO daily for 4 weeks, constituting one cycle. Two cycles of treatment (8 weeks) will be administered followed by a 1-week wash out period during which time patients will be evaluated by the urology oncology team and appropriate surgery will be planned. The wash out period is for drug to be eliminated prior to surgery, to avoid bleeding/wound healing effects. This includes partial nephrectomy or radical nephrectomy. Following surgery, patients with no evidence of disease will have active surveillance. Patients who continue to have disease following surgery will receive further systemic treatment for metastatic disease.

ELIGIBILITY:
INCLUSION CRITERIA Inclusion criteria

* Histologically confirmed locally advanced or metastatic renal cell carcinoma, clear cell histology that can be considered for partial or complete nephrectomy.

  - Locally advanced disease is defined as follows:
  * Adjacent organs (T4) or vascular invasion (Level III/ IV / IVC thrombus)
  * Bulky lymphadenopathy encasing renal or great vessels
* cT1b-T2a Grade (G) 4, cT2b G3/4, c T3-cT4 any grade and any cT with cN1 or M1 disease
* Written and voluntary informed consent.
* Renal function (creatinine level within normal institutional limit, or creatinine clearance >30 mL/min/1.73 m2 for patients with creatinine levels above institutional normal, calculated using the Cockcroft-Gault formula).
* AST/ALT <2.5 X institutional upper limit of normal
* Adequate hematological lab values including:
* Absolute Neutrophil count (ANC) ≥ 1.0 x 109/L
* Platelets ≥ 100 x 109/L
* Hemoglobin ≥ 8.0 g/dL
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 (fully active, able to carry on all pre-disease performance without restriction), 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, such as light housework or office work) or 2 (Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours).
* Age of at least 18 years.
* Life expectancy of 12 weeks or more.
* Measurable disease per RECIST criteria.
* Ejection fraction (EF) ≥ 45%
* Female patients of childbearing potential, as defined in this protocol, must have a negative urine or serum pregnancy test within 72 hours prior to taking the first dose of trial treatment. If the urine test is positive or cannot be confirmed as negative then a serum test is required which must be negative for the patient to enroll. Women of childbearing potential (WOCBP) must be willing to use 2 medically acceptable methods of contraceptive from Day 1 through 120 days after the last dose of trial treatment. The 2 medically acceptable birth control methods can be either 2 barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), copper intrauterine device, sponge, or spermicide as per local regulations or guidelines. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).
* Male patients of childbearing potential, as described in this protocol, must agree to use an adequate method of contraception from Day 1 through 120 days after the last dose of trial treatment.
* Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

EXCLUSION CRITERIA

* Any other cancer from which the patient has been disease-free for less than 3 years (except treated and cured basal-cell or squamous-cell skin cancer, superficial bladder cancer, or treated carcinoma in situ of the cervix, breast, or bladder and treated localized prostate cancer with undetectable PSA for 2 years).
* Symptomatic untreated metastases in the central nervous system.
* Subject that is pregnant or lactating.
* Pre-existing uncontrolled hypertension defined as >140/90 mm Hg with medication.
* Known HIV or acquired immunodeficiency syndrome-related disease.
* Prolongation of QTc interval (>480 ms). QTc interval per Bazett formula.
* Uncontrolled diabetes [fasting glucose >1.5 × upper limit of normal (ULN)] (it will be acceptable if labs were done non-fasting and met the fasting requirement (meaning glucose < 1.5 ULN).
* Fasting total cholesterol >300 mg/dL and fasting triglyceride levels >2.5 × ULN (it will be acceptable if labs were done non-fasting and met the fasting requirement (meaning total cholesterol <300 mg/dL and triglyceride levels < 2.5 × ULN.
* Proteinuria (defined by urine protein/creatinine ratio (UPC) >2.0 if urinalysis protein is >2+)
* Significant cardiovascular impairment: History of (a) congestive heart failure greater than New York Heart association (NYHA) Class II, (b) unstable angina, (c) myocardial infarction (d) stroke, or (e) cardiac arrhythmia associated with hemodynamic instability within 6 months of the first dose of study drugs.
* Known history of active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] RNA detected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Surgical complications as assessed by Clavien-Dindo classification system | Assessment will be completed at the first post-operative visit within 4-6 weeks after surgery.
  To determine whether there is increased surgical morbidity with lenvatinib and everolimus prior to nephrectomy as assessed by Clavien complications.

SECONDARY OUTCOMES:
Treatment related adverse events as assessed by CTCAE criteria, version 4.03 | First treatment through 5 years after Cycle 1, Day 1 or death.
  To assess whether patients will tolerate the combination of lenvatinib and everolimus prior to surgery with same rate of toxicities as seen in prior Phase II clinical trials.
Changes in overall response rate as assessed by RECIST 1.1 | Screening (within 14 days of Day 1) and pre-surgery (week 9-10). 1) If metastatic disease followup monthly or 2) if no evidence of disease followup every three months until five years or death.
  Response and progression will be evaluated using RECIST 1.1. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the criteria. Imaging includes conventional computed tomography (CT) and/or magnetic resonance imagining (MRI), bone scan, and positron emission tomography-computed tomography (PET-CT)
Comparison of surgical outcomes to historical controls | Within two years following the last study participant's surgery
  Review estimated blood loss, blood transfusion, operative time, adjacent organ injury, and postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Yousef Zakharia, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No